CLINICAL TRIAL: NCT00783159
Title: The Effect of Different Training Modalities and Vitamin D Supplementation on Functionality in Prefrail Elderly Persons
Brief Title: Fit in the Aged by Professional Training
Acronym: FiAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Klinikum Nürnberg (Other); Institute of Biomedicine of Aging (Unknown); University of Erlangen-Nürnberg (Other); Institute of Sport Science and Sport (Unknown); Robert Bosch Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32.5.8051.0113.0
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Frailty; Sarcopenia
Keywords: Muscle power; Frailty; Exercise; Vitamin D
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Training I
  Interventions: Procedure: Power Training
- B (Experimental): Training II
  Interventions: Procedure: Strength Training
- C (Active Comparator): Control
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Power Training — Power training, Vitamin D substitution
  Arms: A
Procedure: Strength Training — Strength training, Vitamin D substitution
  Arms: B
Other: Control — Vitamin D substitution, Lifestyle consultation
  Arms: C

SUMMARY:
This intervention study tests training methods to stabilize or improve functionality in the high risk group of prefrail elderly persons.

DETAILED DESCRIPTION:
This study aims at the improvement of muscular function by physical exercise in prefrail elderly persons. Prefrail participants are recruited according to the frailty score of Fried. Taking into account, that vitamin D supplementation reduces falls and improves muscle strength in older people, all participants are supplemented by vitamin D. Two different training methods are tested.

After a run-in period of supplementation of vitamin D for two months, participants will be randomized into three different equally sized groups (n=25): Group A will receive power training. Group B will have progressive strength training. Group C will serve as a control group. They will receive a consultation about leading a healthy life with special attention being paid to nutrition and physical activity. The intervention period lasts for 12 weeks. The 60 minutes training sessions will be held two times a week by members of the Institute of Sport Science and Sports of the University of Erlangen-Nuremberg. Follow-up visits are scheduled three and six months after intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Prefrailty according to the frailty score of Fried

Exclusion Criteria:

* Sarcoidosis
* Nephrolithiasis
* Plasmacytoma
* COPD
* Inflammatory bowel disease
* Rheumatoid arthritis
* History of cancer
* Instable heart disease
* Depression (GDS>=6)
* Dementia (MMSE<=24)
* BMI>35kg/m²
* Current attendance of muscle training
* Medication: immunosuppressive drugs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Short physical performance battery | 3 months after intervention

SECONDARY OUTCOMES:
Muscle strength and muscle power | 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cornel C. Sieber, Prof. Dr., Principal Investigator — University of Erlangen-Nürnberg; Klaus Pfeifer, Prof. Dr., Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Institute of Biomedicine of Aging, Nuremberg, Germany

REFERENCES:
- [Derived] Rippl M, Bidlingmaier M, Deissler L, Martini S, Mueller K, Schluessel S, Schmidmaier R, Schweizer JROL, Tausendfreund O, Welscher L, Drey M. Strength but not power training increases soluble alpha klotho levels in pre-frail older adults. Exp Gerontol. 2026 Jan;213:113002. doi: 10.1016/j.exger.2025.113002. Epub 2025 Dec 13. PMID 41397660
- [Derived] Schaupp A, Bidlingmaier M, Martini S, Reincke M, Schluessel S, Schmidmaier R, Drey M. Resistance training-induced improvement in physical function is not associated to changes in endocrine somatotropic activity in prefrail older adults. Arch Gerontol Geriatr. 2022 Nov-Dec;103:104792. doi: 10.1016/j.archger.2022.104792. Epub 2022 Aug 14. PMID 36037722
- [Derived] Zech A, Drey M, Freiberger E, Hentschke C, Bauer JM, Sieber CC, Pfeifer K. Residual effects of muscle strength and muscle power training and detraining on physical function in community-dwelling prefrail older adults: a randomized controlled trial. BMC Geriatr. 2012 Nov 7;12:68. doi: 10.1186/1471-2318-12-68. PMID 23134737
- [Derived] Drey M, Zech A, Freiberger E, Bertsch T, Uter W, Sieber CC, Pfeifer K, Bauer JM. Effects of strength training versus power training on physical performance in prefrail community-dwelling older adults. Gerontology. 2012;58(3):197-204. doi: 10.1159/000332207. Epub 2011 Nov 3. PMID 22056537